CLINICAL TRIAL: NCT00415129
Title: Safety and Immunogenicity of an Intramuscular Pandemic Influenza Vaccine in Adults and the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GPA02
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; Orthomyxoviridae Infections; Influenza Pandemics; A/H5N1 strain
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group 1 (Experimental): Vaccine with adjuvant
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza virus
- Study Group 2 (Experimental): Vaccine without adjuvant
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza virus

INTERVENTIONS:
Biological: A/H5N1 inactivated, split-virion influenza virus — 0.5mL, Intramuscular
  Arms: Study Group 1
Biological: A/H5N1 inactivated, split-virion influenza virus — 0.5mL, Intramuscular
  Arms: Study Group 2

SUMMARY:
Based on the results from a previous formulation/dosage ranging trial, this phase II multicenter, open trial was designed to determine the safety and immunogenicity of two vaccine formulation/dosages with and without adjuvant 21 days after each vaccination in adults (18 to 60 years and in the elderly (> 60 years) as required by the European Medicines Agency (EMEA) guideline. The antibody persistence until the booster vaccination at 6 or 12 months will also be evaluated.

ELIGIBILITY:
Inclusion Criteria :

* Aged over 18 years on the day of inclusion
* Informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, inability to bear a child or negative urine pregnancy test
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior and at least 4 weeks after to each vaccination.

Exclusion Criteria :

* Systemic hypersensitivity to any component of the vaccine or a life-threatening reaction after previous administration of a vaccine containing the same substances
* Febrile illness (oral temperature ≥ 37.5°C) on the day of inclusion
* Breast-feeding
* Previous vaccination with an avian flu vaccine
* Participation in a clinical trial (drug, device, or medical procedure) within 4 weeks prior to the first vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months or long-term systemic corticosteroid therapy
* Chronic illness that could interfere with trial conduct or completion (e.g. cardiac, renal, diabetes, or auto-immune disorders)
* Current alcohol or drug abuse that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products within the past 3 months
* Any vaccination within 4 weeks prior to the first trial vaccination
* Vaccination planned within 4 weeks after any trial vaccination
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety of an A/H5N1 inactivated, split-virion influenza virus vaccine | 21 Days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (4):
- Belgium (3):
  - Ghent
  - Leuven
  - Wilrijk
- Oxford, United Kingdom

REFERENCES:
- [Derived] Lazarus R, Kelly S, Snape MD, Vandermeulen C, Voysey M, Hoppenbrouwers K, Hens A, Van Damme P, Pepin S, Leroux-Roels I, Leroux-Roels G, Pollard AJ. Antibody Persistence and Booster Responses to Split-Virion H5N1 Avian Influenza Vaccine in Young and Elderly Adults. PLoS One. 2016 Nov 4;11(11):e0165384. doi: 10.1371/journal.pone.0165384. eCollection 2016. PMID 27814377
- [Derived] Leroux-Roels I, Van der Wielen M, Kafeja F, Vandermeulen C, Lazarus R, Snape MD, John T, Carre C, Nougarede N, Pepin S, Leroux-Roels G, Hoppenbrouwers K, Pollard AJ, Van Damme P. Humoral and cellular immune responses to split-virion H5N1 influenza vaccine in young and elderly adults. Vaccine. 2009 Nov 16;27(49):6918-25. doi: 10.1016/j.vaccine.2009.08.110. Epub 2009 Sep 15. PMID 19761837
- See also: Related Info — http://www.sanofipasteur.com